CLINICAL TRIAL: NCT06193551
Title: Ovitex in Paraesophageal and Large Hiatal Hernia Repair. (OviPHeR)
Brief Title: Ovitex in Paraesophageal and Large Hiatal Hernia Repair
Acronym: OviPHeR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foregut Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TelaBio
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Paraesophageal Hernia; Large Hiatal Hernia
Keywords: paraesophageal hiatal hernia; paraesphageal hernia; hiatal hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm of patients undergoing elective repair of paraesphageal hiatal hernia repair or large hiatal henia repair with implant of Ovitex-LPR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients undergoing a paraesophageal or large (>5 cm) hiatal hernia repair (Other): This is a single arm, open label, nonrandomized study evaluating 100 subjects diagnosed with a paraesophageal or large hiatal hernia planning to undergo surgical repair with the study investigators.
  Interventions: Device: Ovitex LPR

INTERVENTIONS:
Device: Ovitex LPR — Robotic assisted laparoscopic repair of hiatal hernia using permanent sutures with Ovitex mesh as reinforcement.

SUMMARY:
The purpose of the study is to evaluate the success of hiatal hernia repairs in patients with large (>5cm) or paraesophageal hernias when Ovitex LPR mesh used during the repair.

DETAILED DESCRIPTION:
This is an investigator initiated, single site, single arm study investigating the recurrence rate of hiatal hernia and safety using Ovitex LPR in patients undergoing hiatal hernia repair.

Ovitex LPR mesh is a reinforced tissue matrix, comprised of a fine non-absorbable polymer suture interwoven through layers of absorbable biologic material in a "lockstitch" pattern.The biologic material in OviTex, derived from ovine rumen (sheep stomach), serves as the natural building block and is optimized to reduce foreign body response, enable functional tissue remodeling and promote a more natural hernia repair. The interwoven polymer fibers provide additional reinforcement, along with improved handling and load-sharing capability. The permanent polymer fiber (polypropylene) is a standard surgical suture material that is used in hiatal hernia surgery and comprises less than 5% of the final product.

Preop details, quality of life questionnaires and surgery details will be collected along with post op GERD (gastro esophageal reflux disease) quality of life questionnaires and barium swallow esophagrams to objectively examine recurrence of hiatal hernia at 1, 3, and 5 years post op. Data will be carefully collected and reviewed for discrepancies and verified with source prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 year old with PEH and appropriate surgical indication for repair

Exclusion Criteria:

* Under 22 years of age.
* In need of an emergency procedure.
* Currently being treated with another investigational drug or device.
* Have had prior gastric or esophageal surgery.
* Have had any previous intervention for GERD.
* Are suspected or confirmed to have esophageal or gastric cancer.
* Have a Body Mass Index (BMI) greater than 45.
* Cannot understand trial requirements or are unable to comply with follow-up schedule.
* Are pregnant, nursing, or plan to become pregnant.
* Have a mental health disorder that would interfere with your ability to follow study instructions.
* Have suspected or known allergies to Ovitex
* Have an illness that may cause you to be unable to meet the protocol requirements or is associated with shortened life expectancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Hiatal Hernia Recurrence as assessed by barium swallow demonstrating axial hernia >2 cm | 5 years
  Assess recurrence rates by objective measures when Ovitex LPR permanent polypropylene polymer reinforcement (Ovitex LPR) is placed during robotic-assisted repair of paraesophageal and large (> 5cm) hiatal hernias (henceforth PEH) using recurrence rate measurements defined as > 2cm axial hernia by Barium Swallow or endoscopy, if available

SECONDARY OUTCOMES:
Number of participants with treatment related mesh erosions as assessed by study quality of life questionnaire leading to endoscopy | 5 years
  Assess the safety of using polypropylene support related to potential erosion as assessed by presence of symptoms using study quality of life questionnaire leading to endoscopy demonstrating mesh erosion

CONTACTS AND LOCATIONS:
Overall Officials: Kate Freeman, MSN, Study Director — Foregut Research Foundation
Locations (1):
- Institute of Esophageal and Reflux Surgery, Lone Tree, Colorado, United States